CLINICAL TRIAL: NCT07305077
Title: One-Minute Preceptor to Improve Bedside Teaching: a Cluster Randomized Trial in Residents
Brief Title: One-Minute Preceptor to Improve Bedside Teaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1925/QĐ-ĐHYDCT/07
Record Dates: First submitted 2025-11-21; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Clinical Teaching; Bedside Teaching; Medical Education

STUDY DESIGN:
Intervention Model Description: Cluster-randomized by preceptor (n=30 clusters; 15 OMP vs 15 control); outcomes at student level
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMP (Experimental): One-Minute Preceptor training: 90-min workshop + pocket card + coaching + fidelity checklist.
  Interventions: Behavioral: One-Minute Preceptor (OMP)
- Control (No Intervention): Usual bedside teaching; OMP offered after trial completion.

INTERVENTIONS:
Behavioral: One-Minute Preceptor (OMP) — Faculty development workshop (90 min), pocket card, coaching, audit with OMP 5-step fidelity checklist.
  Other Names: OMP
  Arms: OMP

SUMMARY:
Intervention Model: Parallel Assignment

Model Description: Cluster-randomized by preceptor (30 clusters; 15 OMP/15 control). Outcomes at student level; 15 students per cluster.

Adequate OMP exposure is defined a priori as ≥2 structured OMP feedback encounters (≥5 minutes each) delivered across ≥2 separate weeks of the rotation.

Masking: Outcomes Assessor

ELIGIBILITY:
Inclusion Criteria:

* A. Student participants (outcome level):

Aged ≥18 years at enrollment.

Enrolled Year 4-medical students assigned to one of the participating preceptor-led bedside teaching groups during the study period.

Expected to attend the rotation for 8-12 weeks (or the site's standard rotation length).

Able to provide informed consent (and agree to be observed/assessed via mini-CEX).

- B. Preceptor clusters (randomized units):

Resident physicians serving as bedside teaching preceptors in participating departments.

Will supervise approximately 15 students during the study period.

Agree not to cross over to teach students in the opposite trial arm during the trial period.

Able to attend OMP training and permit fidelity observation (checklist) if allocated to the intervention.

Exclusion Criteria:

* A. Student participants:

Prior exposure to formal OMP-based teaching within the past 6 months in the same department.

Not expected to remain on the rotation long enough to be assessed (e.g., planned absence >2 weeks or early withdrawal).

Declines or withdraws informed consent.

Severe communication barrier that precludes valid assessment (e.g., language barrier without support).

- B. Preceptor clusters:

Formal OMP training within the past 12 months (to avoid contamination), or role as an OMP trainer for other faculty during the study period.

Planned cross-coverage that would result in teaching students from both arms during the trial period.

Anticipated extended leave making fidelity and outcome assessments infeasible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Mini-Clinical Evaluation Exercise (mini-CEX) Total Score | 8 - 12 weeks
  Total score on the mini-CEX, ranging from 1 to 5. Higher scores indicate better bedside teaching performance as rated by student participants. Measure Type: Continuous.

SECONDARY OUTCOMES:
Student Satisfaction Score | 8-12 weeks
  Description: Student satisfaction with bedside teaching will be measured using a Likert-scale questionnaire specifically developed for this study. The total score ranges from 1 to 5, where higher scores indicate greater satisfaction with the teaching encounter.
  Measure Type: Continuous. Unit of Measure: Score (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Quang C Ngo, Study Chair — Can Tho University Medicine and Pharmacy
Locations (1):
- Can Tho Children Hospital, Can Tho, Province, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided